CLINICAL TRIAL: NCT04032197
Title: A Trial Investigating the Effect of Semaglutide on Atherosclerosis in Patients With Cardiovascular Disease and Type 2 Diabetes
Brief Title: A Research Study of How Semaglutide Works in People With Disease Affecting the Heart and/or Blood Vessels and Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9535-4430; U1111-1215-4058 (Other: World Health Organization (WHO)); 2018-002289-38 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-07-22; First posted 2019-07-25 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Semaglutide injected once-weekly. Standard dose escalations every 4 weeks will be applied, until the maximum dose of 1.0 mg semaglutide is reached.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Placebo injected once-weekly. Standard dose escalations every 4 weeks will be applied, until the maximum dose of 1.0 mg placebo is reached.
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Subcutaneous (s.c., under the skin) injections for 52 weeks. Participants will remain on their pre-study standard of care treatment (antidiabetic medication and CV medication).
  Arms: Semaglutide
Drug: Placebo (semaglutide) — Subcutaneous (s.c., under the skin) injections for 52 weeks. Participants will remain on their pre-study standard of care treatment (antidiabetic medication and CV medication).
  Arms: Placebo

SUMMARY:
This study looks into how the type 2 diabetes medicine, semaglutide, can prevent risk of heart disease complications and stroke. Participants will either get semaglutide or placebo ("dummy" medicine) - which treatment is decided by chance. Semaglutide is a new medicine to treat type 2 diabetes and can be prescribed by doctors in some countries. The study medicine will be in a pen, and must be injected with a needle in the stomach, thigh or upper arm once a week. The study will last for 57-63 weeks. Participants will have 10 clinic visits with the study doctor, 5 visits to the specialised clinic for imaging and at least 1 phone contact. Participants' health will be monitored carefully and blood samples will therefore be taken at the clinic visits. Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age above or equal to 50 years at the time of signing informed consent
* Body mass index equal to or less than 39.9 kg/m^2
* Diagnosed with type 2 diabetes 180 daysor more prior to the day of the first screening visit
* HbA1c 6.0% - 9.0% (42-75 mmol/mol) (both inclusive)
* Established cardiovascular disease

Exclusion Criteria:

* Hospitalisation for unstable angina pectoris or transient ischaemic attack within 90 days prior to the day of the first screening visit
* Planned coronary, carotid or peripheral artery revascularisation.
* Presently classified as being in New York Heart Association (NYHA) equal to or above Class III
* Treatment with glucagon-like peptide-1 receptor agonists (GLP-1 RAs) or systemic anti-inflammatory drugs within 90 days prior to the first screening visit. Stable treatment with acetylsalicylic acid for prevention of cardiovascular events and occasional use of propionic acid derivatives drugs (e.g. ibuprofen) is allowed

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Change in maximum target-to-background ratio (TBR) for 18F-fluorodeoxyglucose (FDG) in the carotid arteries | From baseline (from 41 days before randomisation) to week 26
  Ratio

SECONDARY OUTCOMES:
Change in maximum target-to-background ratio (TBR) for 68Ga-DOTATATE in the carotid arteries | From baseline (from 40 days before randomisation) to week 26
  Ratio
Change in total wall volume of the most diseased carotid artery | From baseline (from 41 days before randomisation) to week 52
  mm3
Change in lipid rich necrotic core (LRNC) volume of the atherosclerotic plaque in the most diseased carotid artery | From baseline (from 41 days before randomisation) to week 52
  mm3
Change in average fibrous cap thickness (FCT) of the atherosclerotic plaque in the most diseased carotid artery | From baseline (from 41 days before randomisation) to week 52
  mm

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (4):
- Clinical Trials Unit / Center for Medical Research, Graz, Austria
- Steno Diabetes Center Copenhagen, Herlev, Denmark
- Sweden (2):
  - Karolinska Universitetssjukhuset Solna,FOU Tema Hjärta Kärl, Stockholm
  - CTC Clinical Trial Consultants AB, Uppsala, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] James S, Christoffersen AD, David JP, Hacker M, Jensen MDRJ, Mellbin L, Pieber TR, Ripa RS, Rossing P, Svehlikova E, Kjaer A. Effect of once-weekly subcutaneous semaglutide on arterial inflammation in people with type 2 diabetes and cardiovascular disease using PET-MRI: Primary results of a randomized, double-blind, placebo-controlled trial. Am Heart J. 2025 Nov;289:17-27. doi: 10.1016/j.ahj.2025.05.001. Epub 2025 May 7. PMID 40345413